CLINICAL TRIAL: NCT02001792
Title: Patient Positioning During Colonoscopy: Effects on Safety and Diagnostic Outcome
Acronym: PACSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PatPo2012
Record Dates: First submitted 2012-04-14; First posted 2013-12-05 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Sedation Problems; Breathing Complications
Keywords: sedation; endoscopy; patient positioning; hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controll group (Sham Comparator): Patients lying in a supine position during colonoscopy
  Interventions: Device: pulse oximeter
- Intervention (Active Comparator): Patients lying in a left lateral position during colonoscopy
  Interventions: Procedure: Position the patient during colonoscopy; Device: pulse oximeter

INTERVENTIONS:
Procedure: Position the patient during colonoscopy — Position the patient either in a left lateral position during colonoscopy
  Arms: Intervention
Device: pulse oximeter

SUMMARY:
The purpose of this study is to determine the effects of patient positioning during colonoscopy on patient safety and diagnostic outcome.

DETAILED DESCRIPTION:
Sedative drugs are widely-used during endoscopic procedures. The administration of these drugs contain the potential hazard of breathing and cardiac complications. Moreover it is well-known that the dorsal position is in some ways associated to breathing problems while patients are asleep. We assume this also to be true related to short anesthesia during colonoscopy. Patient positioning may therefore have a positive effect on the safety during colonoscopy by reducing the absolute time that sedated patients spend in a supine position. We compiled a randomized trial which compares the appearance of breathing and cardiovascular complications by performing colonoscopy either in a dorsal or in a left lateral position.

ELIGIBILITY:
Inclusion Criteria:

* colonoscopy indicated

Exclusion Criteria:

* patient denies sedation
* prior saturation < 90%
* prior heart rate < 50 bpm
* prior blood pressure < 90 mmHg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
frequency of breathing and cardiac problems (decrease of saturation, hypotension, bradycardia) during colonoscopy | participants will be followed for the duration of colonoscopy during hospital stay an expected average of 1 hour
  saturation and heart rate will be measured continuously, blood pressure will be measures all 3 minutes

SECONDARY OUTCOMES:
Adenoma detection rate | 1 day
  Adenoma detection rate between the two arms will be compared at the end of the investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — Departmet for Internal Medicine and Gastroenterology, Technical University Munich, Germany; Stefan von Delius, PD MD, Study Director — Departmet for Internal Medicine and Gastroenterology, Technical University Munich, Germany
Locations (2):
- Germany (2):
  - Endoscopy Section, Department for Internal Medicine and Gastroenterology, Technical University Munich, Munich, Bavaria
  - Krankenhaus Prien, Prien am Chiemsee, Bavaria

REFERENCES:
- [Derived] Klare P, Huth R, Haller B, Huth M, Weber A, Schlag C, Reindl W, Schmid RM, von Delius S. Patient position and hypoxemia during propofol sedation for colonoscopy: a randomized trial. Endoscopy. 2015 Dec;47(12):1159-66. doi: 10.1055/s-0034-1392329. Epub 2015 Jun 30. PMID 26126161